CLINICAL TRIAL: NCT01969370
Title: NCGENES: North Carolina Clinical Genomic Evaluation by NextGen Exome Sequencing
Acronym: NCGENES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, James Evans, MD, PhD, Clinical Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11-1865; U01HG006487 (NIH)
Record Dates: First submitted 2013-10-16; First posted 2013-10-25 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cancer; Cardiovascular Disease; Neurologic Dysfunction; Congenital Abnormalities; Hearing Loss
Keywords: Cancer; Cardiovascular disease; Neurodegenerative disease; Neurodevelopmental disease; Dysmorphology; Hearing loss; Other conditions, including ophthalmic conditions
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Neurologic Manifestations; Congenital Abnormalities; Hearing Loss; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Option to request non-medically actionable incidental information (after receiving education about them)
  Interventions: Behavioral: Experimental
- Control (No Intervention): No option to request non-medically actionable incidental information

INTERVENTIONS:
Behavioral: Experimental — Option to request non-medically actionable incidental information (after receiving education about them)
  Arms: Experimental

SUMMARY:
This study is part of a larger consortium project investigating the validity and best use of next-generation sequencing (in particular, whole exome sequencing, or WES) in clinical care. This sub-project is investigating benefits and harms of providing WES diagnostic and different types of incidental findings to adult patients and parents of pediatric patients who undergo WES because they have symptoms suggesting genetic disease.

DETAILED DESCRIPTION:
This study is part of a larger consortium project investigating the validity and best use of next-generation sequencing (in particular, whole exome sequencing, or WES) in clinical care. Participants are patients who were either seen in the University of North Carolina Cancer and Adult Genetics Clinic or referred to the study by their physician. They will be approached by their physician or a genetic counselor for recruitment. Once enrolled, a clinical geneticist or genetic counselor will obtain consent and collect blood samples to be analyzed using WES. Results may include information related to a diagnosis and incidental information. Medically actionable incidental findings will be CLIA (Clinical Laboratory Improvement Amendments)-certified and returned to participants in a routine genetic counseling session, along with diagnostic findings. Eligible adult participants will be randomized to have the opportunity to choose to get certain types of non-medically actionable incidental findings, as well. Their decisions will be investigated, as will psychosocial and behavioral responses to sequencing and receiving sequencing information. This is a longitudinal, mixed methods study (i.e., multiple assessments pre- and post-return of results, with both quantitative and qualitative methods used to gather data). Because only the quantitative component of the study uses randomization, only measures and procedures associated with that component are described here.

ELIGIBILITY:
- To receive whole exome sequencing in the study, adult or child patients must have a significant chance of having a genetic disorder, as determined by experts on the study team using criteria that depend on the genetic disorder in question. Representative criteria are listed below and will be considered together to determine whether patterns indicate a likely genetic etiology.

Cancer

* Age of diagnosis
* Presence of bilateral (or multiple) cancers
* Diagnosis of a rare type of cancer
* Details of the family history

Cardiovascular Conditions

* Certain clinical findings, such as prolonged QT interval on electrocardiogram.
* Presence of hypertrophic cardiomyopathy or aortic aneurysm
* Age of diagnosis
* Presence of family history

Pediatric neurodevelopmental disorders

* Specific brain structural brain abnormalities
* Presence of certain seizure types
* Dysmorphic features

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2012-08; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Extent of test-specific distress 2 weeks after return of results | 2 weeks after return of diagnostic results; for adult patient participants who are eligible and who request them, 2 weeks after return of non-medically actionable incidental results
  Measured with an adapted version of the multidimensional impact of testing scale (MICRA)

SECONDARY OUTCOMES:
Change in test-specific distress at 3 and 6 months after return of results | Adult patient participants: change from 2 weeks after return of diagnostic results to 3 months and 6 months after return of diagnostic results
  Measure is an adapted version of the multidimensional impact of testing scale MICRA)
Extent of communication of test results with other people | 2 weeks after return of diagnostic results
  Motivations of communications will also be assessed and examined for descriptive analyses.
Extent of information seeking | 2 weeks after consent (T1) and change from T1 to 2 weeks after return of diagnostic results
  Participants will answer questions about the extent to which they sought information about whole exome sequencing and results it produces. Questions also ask about sources of that information (e.g., the Internet, doctors) to provide descriptive data about how participants get information.
Extent of Decision Regret 2 weeks after consent | All participants: 2 wks after consent (T1)
Extent of Decision Regret 2 weeks after return of results | All participants: 2 wks after return of diagnostic (dx) results and, for eligible adults who request them, return of incidental results
  Also administered 2 wks after return of non-medically actionable incidental results for eligible adult patient participants who request them.
Change in decision regret | For all participants: Change from post-consent to post-return of results; Additional for adults: change at 3 and 6 months after return of dx results
Extent of Healthcare Utilization 2 weeks after consent | All participants: 2 wks after consent (T1)
Extent of Healthcare Utilization 2 weeks after return of results | All participants: 22 wks after return of diagnostic (dx) results
Change in Healthcare Utilization | All participants: Change in utilization from post-consent to post-return of results; Additional for adult patients: Change at 3 and 6 months after return of dx results
Enactment of health-related lifestyle behaviors 2 weeks after consent | Adult participants: 2 wks after consent (T1)
  Behaviors include those related to diet, physical activity, smoking, drinking, and substance use.
Enactment of health-related lifestyle behaviors 2 weeks after return of results | Adult participants: 2 wks after return of diagnostic (dx) results
  Behaviors include those related to diet, physical activity, smoking, drinking, and substance use.
Change in enactment of health-related lifestyle behaviors | Adult participants: Change in behaviors from 2 wks after consent (T1) to 2 wks, 3 months, and 6 months after return of dx results
  Behaviors include those related to diet, physical activity, smoking, drinking, and substance use.
Extent of psychological distress 2 weeks after consent | All participants: 2 wks after consent
  Symptoms of depression and anxiety measured with the Hospital Anxiety and Depression Scale
Extent of psychological distress 2 weeks after return of results | All participants: 2 wks after return of diagnostic (dx) results
  Symptoms of depression and anxiety measured with the Hospital Anxiety and Depression Scale
Change in extent of psychological distress | All participants: Change from 2 wks after consent (T1) to 2 wks after return of diagnostic (dx) results; Additional for adult patients: Change at 3 and 6 months after return of dx results
  Symptoms of depression and anxiety measured with the Hospital Anxiety and Depression Scale
Extent of health-related Quality of Life 2 weeks after consent | All participants: 2 wks after consent (T1)
  Measured with the Medical Outcomes Study Short Form-12
Extent of health-related Quality of Life 2 weeks after return of results | All participants: 2 wks after return of diagnostic results
  Measured with the Medical Outcomes Study Short Form-12
Change in extent of health-related Quality of Life | All participants: Change from 2 wks after consent to 2 weeks after return of diagnostic results
  Measured with the Medical Outcomes Study Short Form-12

CONTACTS AND LOCATIONS:
Overall Officials: James P Evans, MD, Ph.D, Principal Investigator — University of North Carolina, Chapel Hill; Gail Henderson, Ph.D, Principal Investigator — University of North Carolina; Jonathan S Berg, MD, Ph.D, Principal Investigator — University of North Carolina; Christine Rini, Ph.D, Study Director — University of North Carolina
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw genotype calls from whole exome sequencing are shared with the database of Genotypes and Phenotypes (dbGaP). Other participant demographic variables include: age of onset, birthplace, sex, race, education level, age.
  Data is uploaded in batches to the dbGaP website. Currently, the data for 403 participants who have consented for release of their data is available on the dbGaP website.
  To access data, users must request authorized access by submitting a Data Use Agreement certified by their institution. This is reviewed by the DbGaP Data Access Committee for approval prior to accessing study data.
  All data that is submitted to dbGaP, including individual participant data, is anonymous.

REFERENCES:
- [Derived] Rini C, Roche MI, Lin FC, Foreman AKM, Khan CM, Griesemer I, Waltz M, Lee K, O'Daniel JM, Evans JP, Berg JS, Henderson GE. Burden or benefit? Effects of providing education about and the option to request additional genomic findings from diagnostic exome sequencing: A randomized controlled trial. Patient Educ Couns. 2021 Dec;104(12):2989-2998. doi: 10.1016/j.pec.2021.04.026. Epub 2021 Apr 29. PMID 33966955